CLINICAL TRIAL: NCT02977000
Title: Department of Neonatology, Children's Hospital of Zhengzhou
Brief Title: Oral Propranolol Improve Retinopathy of Prematurity Outcomes in Very Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huiqing Sun (Other)
Responsible Party: Sponsor-Investigator, Huiqing Sun, Department of Neonatology, Zhengzhou Children's Hospital, China
Organization: Zhengzhou Children's Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROP-PROP
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propranolol (Experimental): Propranolol was administered orally as a dose of 1.5 mg/kg.d divided q8h. investigators used powdered drug, dissolved in 5% dextrose. The treatment was continued until complete development of retinal vascularization, although administration was not permitted for more than 90 days.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Propranolol was administered orally as a dose of 1.5 mg/kg.d divided q8h.investigators used powdered drug, dissolved in 5% dextrose. The treatment was continued until complete development of retinal vascularization, although administration was not permitted for more than 90 days.

SUMMARY:
Retinopathy of prematurity (ROP) is a major cause of blindness and visual impairment in children in both developing and developed countries around the world. ROP is a multifactorial disease characterized by perturbation of normal vascular development in the retina. The pathogenesis of ROP is hypothesized to consist of two distinct phases of which the second phase is characterized by hypoxia-induced up-regulation of vascular endothelial growth factor (VEGF) and retinal neovascularization.

Recent studies have shown a relationship between the β-adrenergic system and angiogenesis. This relationship has been observed in several diseases, like infantile hemangiomas, ROP, and neoplasias. Studies in animal models have shown that norepinephrine stimulates VEGF expression and secretion in retinal cells. In oxygen induced retinopathy, blockage of β-adrenergic receptors (β-AR) can inhibit the angiogenic cascade and interfere with further proliferation of retinal vasculature. Also, angiogenesis seems to be impaired in β-Argene deficient mice, when exposed to hypoxia and other stimuli, but this function is restored after gene therapy.

Assuming in human preterm newborns with ROP that VEGF overexpression and retinal neovascularization in response to hypoxia might involve b-AR activation, we design prospective randomized study to assess the effect of oral propranolol on the progression of early stages of ROP in very low birth weight infants.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is a major cause of blindness and visual impairment in children in both developing and developed countries around the world. ROP is a multifactorial disease characterized by perturbation of normal vascular development in the retina. The pathogenesis of ROP is hypothesized to consist of two distinct phases of which the second phase is characterized by hypoxia-induced up-regulation of vascular endothelial growth factor (VEGF) and retinal neovascularization.

Recent studies have shown a relationship between the β-adrenergic system and angiogenesis. This relationship has been observed in several diseases, like infantile hemangiomas, ROP, and neoplasias. Studies in animal models have shown that norepinephrine stimulates VEGF expression and secretion in retinal cells. In oxygen induced retinopathy, blockage of β-adrenergic receptors (β-AR) can inhibit the angiogenic cascade and interfere with further proliferation of retinal vasculature. Also, angiogenesis seems to be impaired in β-Argene deficient mice, when exposed to hypoxia and other stimuli, but this function is restored after gene therapy.

An association between ROP and infantile hemangiomas was observed over 50 years ago with a higher prevalence of ROP in children with hemangiomas. Studies have also shown that β-AR blockage reduces VEGF levels and favors the regression of infantile hemangiomas. The treatment of choice in threshold stages of ROP is laser photocoagulation and/or intravitreal bevacizumab injections, but management of early stages of ROP, until now has been expectant, with ophthalmologic follow-up but no therapeutic interventions to prevent its progression.

Propranolol is a non-selective β-AR blocker, with equal affinity for β1 and β2 receptors. It has a systemic effect, and acts in different tissues. In vivo models of proliferative retinopathies have shown a strong inhibitory role of β-AR on vascular changes. In particular, β2-AR seems to be the most involved in these responses

. Propranolol has shown to be highly effective in inhibiting both the increase of VEGF expression caused by a hypoxic insult, and the consequent neovascular Response. Studies have shown that propranolol reduces the overproduction of VEGF in oxygen induced retinopathy, but VEGF levels remain unchanged in the normal retina. Assuming in human preterm newborns with ROP that VEGF overexpression and retinal neovascularization in response to hypoxia might involve b-AR activation, we design prospective randomized study to assess the effect of oral propranolol on the progression of early stages of ROP in very low birth weight infants.

Methods:

A randomized controlled trial was performed with preterm newborns with GA <32 weeks of age and Stage 2 ROP without plus in zone II, Although infants were receiving supplemental oxygen, the target range of oxygen saturation was maintained between 91% and 95%. The treated and control newborns are randomized with a 1:1 allocation in blocks of 8 by using a computer random number generator and stratified by center in 2 groups of GA 24-28 and 28-32 weeks; Exclusion criteria included newborns with congenital or acquired cardiovascular anomalies, renal failure or cerebral hemorrhage at enrollment, and newborns with ROP in zone I or at a more advanced stage than Stage 2 without plus in zone II.

With severe adverse effects related to propranolol (severe bradycardia, hypotension, or wheezing), the administration of propranolol was permanently discontinued. If these episodes had been observed within the first 2 days of treatment, these newborns were included into the control group.

All newborns withGA <32 weeks had ophthalmologic evaluations through indirect ophthalmoscopy. When ROP in zone II reached Stage 2 without plus, newborns were enrolled, and ophthalmologic examinations were scheduled weekly or more frequently, according to the severity of ROP. Propranolol was administered orally as a dose of 1.5 mg/kg.d divided q8h. investigators used powdered drug, dissolved in 5% dextrose. The treatment was continued until complete development of retinal vascularization, although administration was not permitted for more than 90 days.

Statistical analyses were performed with the Statistical Software SPSS 17.0. investigators used t tests to assess possible differences in demographic, biochemical, hemodynamic, and respiratory variables between the treated and control newborns. The null hypothesis was accepted with a P > .05. The efficacy of the treatment was evaluated by means of the risk ratio, which is the ratio between the proportion of subjects progressing to more advanced-stage ROP in the propranolol group vs the control group. The relative reduction of risk, which is the reduction percent of events in the treated group vs the control group event rate, was calculated when it was not possible to calculate the risk ratio.

ELIGIBILITY:
Inclusion Criteria:

* preterm newborns with GA <32 weeks of age and Stage 2 ROP without plus in zone II

Exclusion Criteria:

* newborns with congenital or acquired cardiovascular anomalies, renal failure or cerebral hemorrhage at enrollment, and newborns with ROP in zone I or at a more advanced stage than Stage 2 without plus in zone II.

Ages: 24 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The rates of regression of Retinopathy of Prematurity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ligong Hou, MD, Study Chair — Chidren's Hospital of Zhengzhou
Locations (1):
- Propranolol, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No